CLINICAL TRIAL: NCT00978575
Title: Comparison of the Efficacy of Compliant Oral Iron Treatment (FerroDuretter ®) for 3 Months After Discharge Versus Single-dose of Intravenous Iron (Ferinject ®) Before Discharge in Patients With Acute Bleeding From Upper Gastrointestinal Tract. A Double Blinded Randomized Trial
Brief Title: Iron Substitution After Upper Gastro-Intestinal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); Vifor Pharma (Industry)
Responsible Party: Principal Investigator, Palle Bager, Clinical Nurse Specialist, RN, MPH, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Iron Gab
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Gastrointestinal Hemorrhage; Anemia
Keywords: Iron treatment; Upper gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Anemia | interventions — ferric carboxymaltose; serine-ferrosulfate complex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous iron (Active Comparator)
  Interventions: Drug: ferricarboxymaltose
- Oral iron (Active Comparator)
  Interventions: Drug: Ferrosulfate
- Isotonic Sodium and placebo tablets (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ferricarboxymaltose — Single dose of maximum 1000 mg ferricarboxymaltose intravenous
  Other Names: Ferinject
  Arms: Intravenous iron
Drug: Ferrosulfate — 200mg daily for 12 weeks
  Other Names: FerroDuretter
  Arms: Oral iron
Drug: Placebo — 100 mg isotonic sodium and 2 placebo tablets daily
  Arms: Isotonic Sodium and placebo tablets

SUMMARY:
The trial is a double-blind randomized trial designed to examine whether compliant iron therapy (intravenous or oral) for 3 months after discharge increases hemoglobin levels more and faster than no treatment - in patients with acute bleeding from upper gastrointestinal tract. The trial will include 126 patients at Aarhus University Hospital. In addition to efficacy assessment quality of life assessment and health economic calculations between the treatments will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Acute upper gastrointestinal bleeding
* Anemia

Exclusion Criteria:

* Liver disease
* Terminal cancer
* Kidney disease
* variceal bleeding
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
haemoglobin | 13 weeks

SECONDARY OUTCOMES:
Quality of life Health economics | 13 weeks, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Vilstrup, Professor, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Bager P, Dahlerup JF. Randomised clinical trial: oral vs. intravenous iron after upper gastrointestinal haemorrhage--a placebo-controlled study. Aliment Pharmacol Ther. 2014 Jan;39(2):176-87. doi: 10.1111/apt.12556. Epub 2013 Nov 19. PMID 24251969